CLINICAL TRIAL: NCT05445648
Title: Immune Checkpoint Inhibitor in Addition to Transurethral Resection of Bladder Cancer (TUBRT) and Radiation Therapy in Patients With cT2-4aN0M0 Bladder Cancer: a Mono-centre Clinical Study
Brief Title: Comprehensive Bladder Preservation Therapy on Patients With Muscle Invasive Bladder Cancer
Acronym: CBPTMI
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF2022LSK-012
Record Dates: First submitted 2022-06-27; First posted 2022-07-06 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-06

CONDITIONS: Urinary Bladder Neoplasms
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — tislelizumab; Transurethral Resection of Bladder; Radiotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- patients treated with immunotherapy-based bladder preservation therapy (Experimental): Neoadjuvant immunotherapy + TURBT + postoperative adjuvant radiotherapy combined with immunotherapy.
  Interventions: Drug: Tislelizumab Injection; Procedure: Transurethral resection of bladder tumor; Radiation: Adjuvant radiotherapy

INTERVENTIONS:
Drug: Tislelizumab Injection — After patient recruitment, every patient first receives a regimen of tislelizumab injection 200 mg every time , q3w, 4 times in total. Then all patients, if operable, undergo TURBT. The first day after TURBT, patients again start to receives a regimen of tislelizumab Injection 200 mg every time , q3w, 4 times in total. Meanwhile, on the eighth day after TURBT, patients start to receive radiotherapy. The total radiation dosage is 50.4 Gy (patients receive radiotherapy 28 times, dosage being 1.8 Gy every time), with the total radiation dosage on pelvis area being 45 Gy and total radiation dosage on bladder area being 50.4 Gy.
  Other Names: BGB-A317; BeiGene
Procedure: Transurethral resection of bladder tumor — After the initial tislelizumab injection regimen, patients undergo clinical assessment and receive transurethral resection of bladder tumor if operable.
Radiation: Adjuvant radiotherapy — On the eighth day after TURBT, patients start to receive radiotherapy. The total radiation dosage is 50.4 Gy (patients receive radiotherapy 28 times, dosage being 1.8 Gy every time), with the total radiation dosage on pelvis area being 45 Gy and total radiation dosage on bladder area being 50.4 Gy.

SUMMARY:
Nowadays, Immune Checkpoint Inhibitor (ICI) has become one of the new drugs for the treatment of advanced uroepithelial carcinoma. The Food and Drug Administration (FDA) approved ICI for bladder cancer (BC) patients who cannot tolerate cisplatin chemotherapy and whose tumors express programmed cell death protein ligand-1 (PD-L1). However, the efficacy of ICI in bladder preservation therapy for muscular invasive bladder cancer (MIBC) is unknown.

With the progressive clinical confirmation of the efficacy of immunotherapy, ICI has moved from second-line to first-line treatment in the indication of advanced unresectable BC. It even has been used in the neoadjuvant and postoperative adjuvant therapy for MIBC and non-muscle invasive bladder cancer (NMIBC) where Bacillus Calmette-Guérin (BCG) therapy has failed. Available studies have shown that neoadjuvant immunotherapy can achieve a pathological complete response (pCR) of 31%-42% for MIBC, regardless of using a single drug or combination, which is higher than that of neoadjuvant chemotherapy, and the incidence of side effects associated with neoadjuvant immunotherapy is lower than that of neoadjuvant chemotherapy, providing an effective treatment option for cisplatin-intolerant patients.

Studies have shown that radiotherapy leads to immunogenic cell death, which results in the release and presentation of tumor antigens and directs the recruitment and activation of T cells. It also induces increased expression of PD-L1 in tumor cells, which in turn improves the efficacy of immunotherapy. Thus ICI combined with radiotherapy has a synergistic antitumor effect and does not produce serious toxic side effects similar to those associated with chemotherapeutic agents.

This study proposes a novel neoadjuvant immunotherapy-based integrated bladder preservation therapy (neoadjuvant immunotherapy + TURBT + postoperative adjuvant radiotherapy combined with immunotherapy) and investigates the effectiveness and safety of this strategy in bladder preservation treatment strategy.

DETAILED DESCRIPTION:
This study aims to investigate the efficacy and safety of a comprehensive immunotherapy-based bladder preservation treatment strategy (neoadjuvant immunotherapy + TURBT + adjuvant radiation therapy (RT) combined with immunotherapy) by implementing a prospective, single-arm, single-center, open clinical trial.

It aims to: 1) assess pCR (pathological complete remission rate) and pathological stage reduction rate of patients with MIBC after neoadjuvant immunotherapy. 2) assess relative risk factors that have an impact on pathological stage reduction rate and pCR. 3) assess bladder preservation rate of MIBC patients after the immunotherapy-based integrated bladder preservation therapy. 4) assess tumor recurrence-free survival, progression-free survival, and tumor-specific and overall survival rates after treatment. 5) To assess the safety of this treatment. 6) To collect tumor tissues from TURBT and study genetic variations as well as the expression of relevant biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Voluntary participation in this trial, able to provide a written version of informed consent, and able to understand and agree to comply with the requirements of this study.
* BC patients with cT2-T4aN0M0 tumor/ lymph node/ metastasis (TNM) (AJCC 8th edition) staging based on histopathological confirmation by biopsy specimen and CT/MRI assessment.
* ECOG performance status grade less than or equal to 1

Exclusion Criteria:

* Cancer in situ (CIS) confirmed by biopsy pathology.
* Prior treatment with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-cytotoxic T-lymphocyte-associated protein 4(CTLA)-4 antibody or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways (excluding BCG treatment).
* Received other approved systemic anticancer therapy or systemic immunomodulators within 28 days prior to enrollment.
* Severe chronic or active infection requiring systemic antibacterial, antifungal or antiviral therapy within 14 days prior to enrollment
* Received herbal or proprietary Chinese medicine for cancer inhibition within 14 days prior to admission.
* Received live vaccination within 28 days prior to admission.
* Has need for long-term heavy use of hormones or other immunosuppressive drugs.
* Potassium, sodium, or calcium abnormalities affecting treatment, interstitial lung disease, non-infectious pneumonia, or other uncontrolled systemic diseases, including diabetes, hypertension, or active heart disease.
* Patients with chronic hepatitis B, hepatitis B virus carriers, or active hepatitis C.
* Active, known or suspected autoimmune disease requiring systemic therapy.
* Patients with end-stage renal disease (GFR <15 mL/min) or requiring dialysis.
* Other active neoplastic disease.
* Uncontrolled severe physical or mental illness.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Bladder preservation rate within 1 year, % | 1 year after neoadjuvant immunotherapy (Tislelizumab Injection) started
  The percentage of enrolled patients who didn't receive radical cystectomy 1 year after neoadjuvant immunotherapy (Tislelizumab Injection) started
Pathological complete response rate after neoadjuvant immunotherapy, % | right after TURBT and pathological examination of surgical specimen has concluded.
  the percentage of enrolled patients who demonstrated pathological complete response after neoadjuvant immunotherapy, confirmed by pathological results of specimen extracted from TURBT.

SECONDARY OUTCOMES:
Overall survival time, day | from the start of neoadjuvant immunotherapy to 1) death of the patients by any cause; 2) the end of followup if patients are still alive by that time; 3) last follow up date if patients are lost, whichever comes first, assessed up to 156 weeks
  the time from the start of neoadjuvant immunotherapy to 1) death of the patients by any cause; 2) the end of followup if patients are still alive by that time; 3) last follow up date if patients are lost, whichever comes first
Adverse event | from the start of neoadjuvant immunotherapy to the last followup check, assessed up to 156 weeks
  all adverse events ever occurred to enrolled patients from the start of neoadjuvant immunotherapy to the last followup check, coded by MedDra. The severity of adverse effect will be evaluated by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Jinhai Fan, MD, Principal Investigator — First affiliated hospital of Xian jiaotong university
Locations (1):
- First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi, China